CLINICAL TRIAL: NCT01277757
Title: Phase II Trial of AKT Inhibitor MK2206 in Patients With Advanced Breast Cancer Who Have Tumors With a PIK3CA Mutation, or an AKT Mutation, and/or PTEN Loss/PTEN Mutation
Brief Title: Akt Inhibitor MK2206 in Treating Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02892; NCI-2012-02892 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2010-0242; CDR0000694003; 2010-0242 (Other: M D Anderson Cancer Center); 8732 (Other: CTEP); N01CM00039 (NIH); N01CM62202 (NIH); P30CA016672 (NIH); U01CA062490 (NIH)
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Recurrent Breast Carcinoma; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — MK 2206

ARMS (1):
- Treatment (Akt inhibitor MK-2206) (Experimental): Akt Inhibitor MK-2206 mg orally once a week on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given orally (PO) weekly, starting (dose 0) at 200 mg
  Other Names: MK2206
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well Akt inhibitor MK2206 works in treating patients with breast cancer cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment. Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether v-akt murine thymoma viral oncogene (Akt) inhibitor MK2206 achieves objective tumor responses (complete response [CR], partial response [PR]) in advanced breast cancer patients who have a phosphoinositide-3-kinase, catalytic, alpha polypeptide (PIK3CA) or Akt mutation and/or phosphatase and tensin homolog (PTEN) loss or mutation.

SECONDARY OBJECTIVES:

I. To determine the 6 month progression-free survival on MK2206. II. To determine baseline molecular markers that may predict clinical outcome. III. To determine pharmacodynamic markers in blood and tumor tissue that may predict a decrease in proliferation-related Ki-67 antigen (Ki-67) and clinical outcome.

IV. To determine safety and tolerability of MK2206 in previously treated patients with advanced breast cancer.

V. To determine if decrease in Ki-67 at 2 weeks correlates with anti-tumor effect (CR, PR, or stable disease [SD] > 6 months).

VI. To determine concordance of PIK3CA and PTEN status between primary tumor and distant metastasis.

VII. To determine concordance of PIK3CA status of circulating free deoxyribonucleic acid (DNA) and distant metastasis.

OUTLINE:

Patients receive Akt Inhibitor MK-2206 orally (PO) on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed breast cancer, with diagnosed or suspected metastatic, inoperable locally advanced breast cancer, or inoperable locally recurrent breast cancer
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan
* Patients who have failed to respond to at least one line of systemic therapy are eligible for MK2206 therapy; if the patient has a human epidermal growth factor receptor 2 (HER2) positive tumor, it is expected that they will have received at least one HER2-targeted therapy in the metastatic setting; if the patient has an estrogen receptor positive (ER+) tumor, it is expected that they will have received at least one ER-targeted therapy in the metastatic setting; patients can be enrolled for molecular screening while on another therapy if the patient is interested in MK2206 therapy upon progression
* Archived primary tumor biopsies or surgical specimens, or biopsies of recurrence or metastasis, will be available for PIK3CA/Akt mutational analysis and PTEN analysis; patients with surgical samples, or core/punch biopsies available, will be eligible for testing for PIK3CA/Akt status as well as PTEN testing; the most recent sample will be preferred (i.e. in patients with metastatic disease, metastases samples are preferred over archival primary tumor and in patients with local recurrences a biopsy of the recurrence is preferred over archival primary tumor); NOTE: PIK3CA or Akt mutation status can be determined on fine needle aspirate (FNA) samples, but PTEN status cannot as stroma and endothelial cells are used as internal controls and PTEN testing has not been validated on FNA samples; thus patients with only FNA samples and no tissue blocks available will be considered to be eligible for screening for PIK3CA/Akt mutations and will be enrolled onto the study only if they are found to have PIK3CA mutations or Akt mutations; patients whose tumors have already been tested in the Clinical Laboratory Improvement Amendments (CLIA) environment and have been found to have a PIK3CA mutation or Akt mutation or PTEN loss by immunohistochemistry (IHC) or PTEN mutation will be eligible for treatment; patients whose tumors have been tested in the research environment and found to have a PIK3CA mutation or Akt mutation or PTEN loss or PTEN mutation will have their marker status confirmed in the CLIA environment
* Patients whose tumors have already been tested in the CLIA environment and have been found to have a PIK3CA mutation or Akt mutation or PTEN loss or mutation will be eligible for treatment; patients whose tumors have been tested in the research environment and found to have a PIK3CA mutation or Akt mutation or PTEN loss or mutation will have their marker status confirmed in the CLIA environment.
* Patient will have a tumor suitable for FNA and/or core/punch biopsy for research purposes
* Patient must have Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelets >= 100,000/uL
* Hemoglobin (Hgb) >= 9 g/dL
* Creatinine =< 1.5 X upper limit of normal (ULN)
* Prothrombin time (PT), partial thromboplastin time (PTT) =< 1.2 X ULN
* Total bilirubin =< 1.5 X ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 X ULN
* Patients of childbearing potential must have a negative serum or urine pregnancy test beta-human chorionic gonadotropin (hCG) within 72 hours prior to study registration
* Women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and also for 4 weeks after the end of therapy; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately
* Patient must have completed any systemic therapy regimens and therapeutic radiation a minimum of 21 days prior to initiation of study therapy
* Ability to understand and the willingness to sign a written informed consent document
* >= 6 months life expectancy as documented in patient records

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events to grade 1 or less due to agents administered more than 3 weeks earlier
* Patients may have received prior investigational therapies; however, they not be receiving any other investigational agents concurrent with MK2206; patients must have completed therapy a minimum of 21 days prior to initiation of study therapy
* Patients may not have received treatment with another inhibitor of phosphatidylinositol 3 kinase (PI3K), Akt or mammalian target of rapamycin (mTOR) in the neoadjuvant, adjuvant or metastatic setting with the exception of rapalogs; patients with metastatic breast cancer, who received PI3K/Akt/mTOR inhibitors on short preoperative window trials (treatment for 4 weeks or less), will be eligible if the treatment was over 6 months prior to registration; patients must have completed therapies a minimum of 21 days prior to initiation of study therapy
* Patients with known brain metastases should be excluded from this clinical trial; patients will not undergo pre-treatment imaging of the brain, unless clinically indicated
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK2206 or other agents used in the study
* Patients receiving any medications or substances that are potent inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP 450 3A4) are ineligible; however, patients will be permitted regular dietary consumption of caffeine; glyburide will be allowed for the treatment of hyperglycemia
* Patients with diabetes or in risk for hyperglycemia should not be excluded, but patients with poorly controlled diabetes (glycated hemoglobin [HBA1C] > 8%) should be excluded
* Baseline corrected QT by Fridericia's formula (QTcF) > 450 msec (male) or QTcF >b470 msec (female) will exclude patients from entry on study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Baseline bradycardia related to cardiac disease, or significant bundle branch block
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with MK2206
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients at high risk for coagulopathy
* Liver disease burden greater or equal to 50 percent
* Need for blood or platelet transfusion within one month from baseline laboratory testing as well as within treatment initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Xing Y, Lin NU, Maurer MA, Chen H, Mahvash A, Sahin A, Akcakanat A, Li Y, Abramson V, Litton J, Chavez-MacGregor M, Valero V, Piha-Paul SA, Hong D, Do KA, Tarco E, Riall D, Eterovic AK, Wulf GM, Cantley LC, Mills GB, Doyle LA, Winer E, Hortobagyi GN, Gonzalez-Angulo AM, Meric-Bernstam F. Phase II trial of AKT inhibitor MK-2206 in patients with advanced breast cancer who have tumors with PIK3CA or AKT mutations, and/or PTEN loss/PTEN mutation. Breast Cancer Res. 2019 Jul 5;21(1):78. doi: 10.1186/s13058-019-1154-8. PMID 31277699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 14, 2011 to November 27, 2013. Recruitment done at The University of Texas MD Anderson Cancer Center, Beth-Israel Deaconness, Columbia University Medical Center, Dana Farber Cancer Center and Vanderbilt University.
Pre-assignment Details: Of the 30 participants registered, two were ineligible, not treated therefore excluded from the trial outcomes.
Groups:
- Akt Inhibitor MK-2206: Akt Inhibitor MK-2206 orally once a week on days 1, 8, 15, and 22. Starting dose 200 mg, courses repeat every 28 days.
Period: Overall Study
Arm/Group | Akt Inhibitor MK-2206
Started | 30
Completed | 28
Not Completed | 2
Not completed — Disease Progression | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Two participants were not treated.
Arm/Group | Akt Inhibitor MK-2206
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 52.5 [31 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response Defined Using Response Evaluation Criteria In Solid Tumors (RECIST)
Description: Number of participants with response defined by RECIST version 1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: appearance of one or more new lesions is also considered progressions). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 3 weeks after completion of study treatment, for up to 1 year
Population: Two participants were not treated therefore excluded from study population analysis, another was inevaluable and six others were not analyzable for response.
Measure: Number; unit: participants
Arm/Group | Akt Inhibitor MK-2206
Number analyzed (Participants) | 21
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 1
  Progressive Disease (PD) | 20
  Stable Disease (SD) | 0

2. Primary Outcome: Number of Participants With Objective Response
Description: Only those participants who have measurable disease present at baseline, have received at least four doses of MK2206, and have had their disease re-evaluated will be considered evaluable for response. Response classified according the RECIST definitions, and re-evaluated for response every 12 weeks. (Note: Participants who exhibit objective disease progression prior to receiving four doses of therapy will also be considered evaluable.) In addition to a baseline scan, confirmatory scans should also be obtained 4-6 weeks following initial documentation of objective response, and then revert to scheduled repeat imaging.
Time Frame: 4 weeks following beginning treatment, repeat confirmation 4-6 weeks following response, up to 1 year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Akt Inhibitor MK-2206
Number analyzed (Participants) | 21
participants | 8

3. Secondary Outcome: 6 Month Progression-free Survival (PFS)
Description: Number of participants progression free at 6 months. PFS is defined as the duration of time from start of treatment, or time of progression or death, whichever occurs first. The PFS for this outcome was assessed at 6 months post treatment.
Time Frame: From start of treatment to time of progression or death or six months whichever occurs first, assessed at 6 months
Measure: Number; unit: participants
Arm/Group | Akt Inhibitor MK-2206
Number analyzed (Participants) | 27
participants | 0

4. Secondary Outcome: Median Response Duration
Description: The duration of the response is from the time response is achieved until disease progression is detected. The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented.
  Response re-evaluated every 12 weeks. In addition to a baseline scan, confirmatory scans should also be obtained 4-6 weeks following initial documentation of objective response.
Time Frame: Response assessment 4 weeks from beginning of treatment, response recorded from the start of treatment until disease progression/recurrence, up to 1 year
Population: Two participants were not treated, and one was inevaluable.
Measure: Median (Full Range); unit: months
Arm/Group | Akt Inhibitor MK-2206
Number analyzed (Participants) | 27
months | 5.8 [0.1 to 7.0]

5. Other Pre Specified Outcome: Apoptosis Assessed by Cleaved Caspase-3
Description: Assessment of apoptosis by immunohistochemistry to active caspase-3. Initially, the goal was to look at predictors of response, but the number of responses was not enough to make a determination.
Time Frame: Up to 30 days after completion of study treatment, up to 1 year
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Cell Proliferation as Measured by the Change in Percent Ki-67 Positive Cells
Description: Ki-67 will be scored as % positive cells to determine whether there is a change % Ki-67+ cells before treatment versus after 2 weeks of treatment. Initially, the goal was to look at predictors of response, but the number of responses was not enough to make a determination.
Time Frame: Baseline to 2 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Event collection during each cycle, with a cycle duration being 28 days then followed for 3 weeks after removal from treatment or until death, whichever occurs first, for up to 1 year. Overall collection period: May 2011 to May 2014.
Arm/Group | Akt Inhibitor MK-2206
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 24/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Akt Inhibitor MK-2206 (N=28)
Hematocrit drop (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Akt Inhibitor MK-2206 (N=28)
Examplex (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 2 (4)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 5 (9)
Anorexia (Metabolism and nutrition disorders) | 4 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 5 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (3)
Blood bilirubin increased (Metabolism and nutrition disorders) | 1 (5)
Blurred vision (Eye disorders) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Creatinine increased (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (35)
Dizziness (Nervous system disorders) | 3 (3)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 4 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Edema limbs (General disorders) | 3 (4)
Fatigue (General disorders) | 17 (52)
Fever (General disorders) | 4 (4)
Flu like symptoms (General disorders) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (7)
Hypertension (Vascular disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infections and infestations - (Other) (Infections and infestations) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (15)
Investigations - (Other) (Investigations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 5 (12)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (12)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 10 (30)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - (Other) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Nervous system disorders - (Other) (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Pain of skin (Skin and subcutaneous tissue disorders) | 5 (7)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 6 (16)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Platelet count decreased (Investigations) | 1 (4)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (38)
Scleral disorder (Eye disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (6)
Skin and subcutaneous tissue disorders - (Other) (Skin and subcutaneous tissue disorders) | 3 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Vertigo (Eye disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (11)
Weight loss (Investigations) | 2 (5)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less